CLINICAL TRIAL: NCT00259610
Title: Treatment of Early Aggressive Rheumatoid Arthritis (TEAR)
Acronym: TEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Amgen (Industry); Barr Laboratories (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X031030004; 20040391
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2013-10

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; painful joints; swollen joints
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthralgia | interventions — Methotrexate; Sulfasalazine; Hydroxychloroquine; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): methotrexate (MTX) + etanercept
  Interventions: Drug: methotrexate; Drug: etanercept
- 2 (Active Comparator): methotrexate (MTX) + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
  Interventions: Drug: methotrexate; Drug: sulfasalazine; Drug: hydroxychloroquine
- 3 (Active Comparator): methotrexate (MTX) or MTX + Etanercept
  Interventions: Drug: methotrexate; Drug: etanercept
- 4 (Active Comparator): methotrexate (MTX) or MTX + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
  Interventions: Drug: methotrexate; Drug: sulfasalazine; Drug: hydroxychloroquine

INTERVENTIONS:
Drug: methotrexate — varies
Drug: sulfasalazine — varies
  Arms: 2; 4
Drug: hydroxychloroquine — varies
  Arms: 2; 4
Drug: etanercept — varies
  Arms: 1; 3

SUMMARY:
The purpose of this study is to 1)to determine if it is better to treat all early RA patients with methotrexate in combination with hydroxychloroquine plus sulfasalazine or in combination with etanercept or reserve this treatment for patients who do not appropriately respond to methotrexate alone and 2) to determine which combination of methotrexate therapy is better

DETAILED DESCRIPTION:
The ultimate goal of RA is to eliminate symptoms, restoring the patient to normal physical, social, emotional, and vocational function, and preserving the structure and integrity of joints. While disease modifying anti-rheumatic drugs (DMARDs) have long been the cornerstone of RA therapy, the limitations of DMARDs have become increasingly apparent and investigators continue to gain insight into the pathogenesis of this disease. Recent evidence suggests that treatment earlier in the disease process with more aggressive approaches results in superior long-term outcomes compared to less intensive treatment regimens. Specifically, there is growing interest in the possibility that early "aggressive" treatment with combinations of DMARDs as initial treatment in efforts to potentially reduce the proportion of patients that advance to severe disability.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of RA for less than or equal to 3 years
* Be 18 years of age or older at the time of diagnosis

Exclusion Criteria:

* Pregnant or lactating women
* History of chronic infection, such as hepatitis, pneumonia, or chronic skin infections
* Active TB or evidence of latent TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2004-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Curtis, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Moreland LW, O'Dell JR, Paulus HE, Curtis JR, Bathon JM, St Clair EW, Bridges SL Jr, Zhang J, McVie T, Howard G, van der Heijde D, Cofield SS; TEAR Investigators. A randomized comparative effectiveness study of oral triple therapy versus etanercept plus methotrexate in early aggressive rheumatoid arthritis: the treatment of Early Aggressive Rheumatoid Arthritis Trial. Arthritis Rheum. 2012 Sep;64(9):2824-35. doi: 10.1002/art.34498. PMID 22508468
- [Derived] Charles-Schoeman C, Yin Lee Y, Shahbazian A, Wang X, Elashoff D, Curtis JR, Navarro-Millan I, Yang S, Chen L, Cofield SS, Moreland LW, Paulus H, O'Dell J, Bathon J, Louis Bridges S Jr, Reddy ST. Improvement of High-Density Lipoprotein Function in Patients With Early Rheumatoid Arthritis Treated With Methotrexate Monotherapy or Combination Therapies in a Randomized Controlled Trial. Arthritis Rheumatol. 2017 Jan;69(1):46-57. doi: 10.1002/art.39833. PMID 27483410
- [Derived] Hwang YG, Balasubramani GK, Metes ID, Levesque MC, Bridges SL Jr, Moreland LW. Differential response of serum amyloid A to different therapies in early rheumatoid arthritis and its potential value as a disease activity biomarker. Arthritis Res Ther. 2016 May 17;18(1):108. doi: 10.1186/s13075-016-1009-y. PMID 27188329
- [Derived] Charles-Schoeman C, Wang X, Lee YY, Shahbazian A, Navarro-Millan I, Yang S, Chen L, Cofield SS, Moreland LW, O'Dell J, Bathon JM, Paulus H, Bridges SL Jr, Curtis JR. Association of Triple Therapy With Improvement in Cholesterol Profiles Over Two-Year Followup in the Treatment of Early Aggressive Rheumatoid Arthritis Trial. Arthritis Rheumatol. 2016 Mar;68(3):577-86. doi: 10.1002/art.39502. PMID 26606398
- [Derived] Maska LB, Sayles HR, O'Dell JR, Curtis JR, Bridges SL Jr, Moreland LW, Cofield SS, Mikuls TR. Serum cotinine as a biomarker of tobacco exposure and the association with treatment response in early rheumatoid arthritis. Arthritis Care Res (Hoboken). 2012 Dec;64(12):1804-10. doi: 10.1002/acr.21758. PMID 22730343
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22508468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May 2004 and concluded in January 2007.
Pre-assignment Details: This study had a screening period of 1-3 days, Patients were excluded for various reasons, including, laboratory exclusions, Positive TB test, and Cataract/visual defect.
Groups:
- MTX + Active Etanercept: Methotrexate (MTX)5mg -20mg/qw by mouth(within 12 weeks of entry in study) + etanercept 50mg/qw by injection
- MTX+ Active SSZ +HCQ: methotrexate (MTX)20mg/qw by mouth(within 12 weeks of entry in study) + sulfasalazine (SSZ) 500mg qd - 1000mg 2qd by mouth /hydroxychloroquine (HCQ)200mg 2qd by mouth
- MTX + Placebo Entaneracept: Methotrexate (MTX)5mg -20mg/qw by mouth(within 12 weeks of entry in study) + Etanercept(Placebo) 50mg/qw by injection
- MTX + Placebo SSZ + HCQ(ST): Methotrexate (MTX)5mg -20mg/qw by mouth(within 12 weeks of entry in study) + sulfasalazine (SSZ) 500mg qd - 1000mg 2qd by mouth /hydroxychloroquine (HCQ)200mg 2qd by mouth
Period: Overall Study
Arm/Group | MTX + Active Etanercept | MTX+ Active SSZ +HCQ | MTX + Placebo Entaneracept | MTX + Placebo SSZ + HCQ(ST)
Started | 244 | 132 | 255 | 124
Completed | 168 | 86 | 182 | 81
Not Completed | 76 | 46 | 73 | 43
Not completed — Withdrawal by Subject | 33 | 25 | 29 | 19
Not completed — Lost to Follow-up | 19 | 8 | 18 | 15
Not completed — Physician Decision | 6 | 4 | 7 | 2
Not completed — Death | 1 | 1 | 2 | 0
Not completed — non medical reason | 6 | 2 | 10 | 3
Not completed — Adverse Event | 3 | 4 | 5 | 2
Not completed — Serious Adverse Event | 8 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- MTX + Active Etanercept: Methotrexate (MTX) + etanercept
- MTX+ Active SSZ +HCQ: methotrexate (MTX) + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
- MTX + Placebo Entaneracept: methotrexate (MTX) or MTX + Etanercept
- MTX + Placebo SSZ + HCQ(ST): methotrexate (MTX) or MTX + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
- Total: Total of all reporting groups
Arm/Group | MTX + Active Etanercept | MTX+ Active SSZ +HCQ | MTX + Placebo Entaneracept | MTX + Placebo SSZ + HCQ(ST) | Total
Number analyzed (Participants) | 244 | 132 | 255 | 124 | 755
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 244 | 132 | 255 | 124 | 755
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.4) | 48.8 (12.7) | 48.6 (13.0) | 49.3 (12.0) | 49.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 101 | 176 | 87 | 545
  Male | 63 | 31 | 79 | 37 | 210
Region of Enrollment [Number; unit: participants]
  United States | 244 | 132 | 255 | 124 | 755

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score Erythrocyte Sedimentation Rate(DAS28-ESR)
Description: Outcome measured was the observed-group analysis of the DAS28-ESR between weeks 48 and 102. DAS28 is a calculated scale using a formula that includes the number of tender joints and swollen joints (28 joints maximum). The following is the calculation: DAS28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * GH. The ESR is the rate at which red blood cells sediment in a period of one hour.
  The total range for the DAS28ESR goes from 0.0 to 9.2; this indicates the current activity of the rheumatoid arthritis of a subject. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity.
Time Frame: Change of the Mean of DAS28-ESR between weeks 48 - 102.
Population: The participants that were randomized into this clinical trial and completed the study to year 2, represent the number for analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- MTX + Immediate Etanercept: Methotrexate (MTX) + etanercept
- MTX+ Immediate SSZ +HCQ: methotrexate (MTX) + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
- MTX + Step-up Etanercept: methotrexate (MTX) or MTX + Etanercept
- MTX + Step-up SSZ + HCQ(ST): methotrexate (MTX) or MTX + sulfasalazine (SSZ)/hydroxychloroquine (HCQ)
Arm/Group | MTX + Immediate Etanercept | MTX+ Immediate SSZ +HCQ | MTX + Step-up Etanercept | MTX + Step-up SSZ + HCQ(ST)
Number analyzed (Participants) | 159 | 76 | 166 | 75
Scores on a scale | 3.0 (1.4) | 2.9 (1.5) | 3.1 (1.4) | 2.8 (1.3)

2. Secondary Outcome: Radiographic Disease Progression Between Baseline and Week 102 as Assessed by Van Der Heijde Modified Sharp Scores.
Description: Changes in disease progression between treatment groups will be described by the mean score at two years as assessed after adjustment for the baseline radiographic score. Radiographs were observed of hands, wrists, and feet. The range of scores available for the modified Sharp Score is 0 to 448. The erosion score per joint of the hands can range from 0 to 5. The maximal erosion score for each hand is thus 80, considering the 16 areas for erosions per hand. Joint space narrowing and joint subluxation or luxation are combined in a single score with a range of 0 to 4 with a max score of 60. The erosion score per joint can range from 0 to 10, with each side of the joint independently scored from 0 to 5. The maximal erosion score per foot is thus 60. The joint space narrowing and joint (sub)luxation are combined in a single score with a range of 0 to 4. The maximal narrowing/(sub)luxation score per foot is thus 24.
Time Frame: Year 2, Week 102
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MTX + Immediate Etanercept | MTX+ Immediate SSZ +HCQ | MTX + Step-up Etanercept | MTX + Step-up SSZ + HCQ(ST)
Number analyzed (Participants) | 159 | 76 | 166 | 75
Scores on a scale | 7.0 (16.6) | 7.3 (13.3) | 4.8 (7.2) | 6.2 (8.9)

ADVERSE EVENTS:
Arm/Group | MTX + Active Etanercept | MTX+ Active SSZ +HCQ | MTX + Placebo Entaneracept | MTX + Placebo SSZ + HCQ(ST)
Serious Adverse Events (participants affected / at risk) | 35/244 | 18/132 | 32/255 | 16/124
Other Adverse Events (participants affected / at risk) | 184/244 | 99/132 | 180/255 | 89/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTX + Active Etanercept (N=244) | MTX+ Active SSZ +HCQ (N=132) | MTX + Placebo Entaneracept (N=255) | MTX + Placebo SSZ + HCQ(ST) (N=124)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Arterial Thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial Blockage (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Death (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Anterior Descending Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Other Infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dilated Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea / Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other Infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perforated Bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncopal Episode (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other Infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Elevated LFTs (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Low Hemoglobin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Cerebellar Infarcation w/ Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical Procedure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cancer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis Carini (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Vascular Accident (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Replacement (Surgical and medical procedures) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Joint Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other Infection (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perforated Bowel (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical Procedure (Surgical and medical procedures) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Pulmonary Edema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolus (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischemic Attack (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTX + Active Etanercept (N=244) | MTX+ Active SSZ +HCQ (N=132) | MTX + Placebo Entaneracept (N=255) | MTX + Placebo SSZ + HCQ(ST) (N=124)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 8 (8) | 3 (3) | 7 (7) | 2 (2)
Nose Bleed (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 5 (5) | 1 (1) | 4 (4) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 6 (6) | 1 (1) | 4 (4) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
SHORTNESS OF BREATH (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR HYPERTROPHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EAR CONGESTION/FULLNESS (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
EARACHE/ INFECTION (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
HEARING LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DIABETES (Endocrine disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
HYPO/HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
THYROID ENLARGEMENT/NODULES (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
DECREASED VISION (Eye disorders) | 2 (2) | 4 (4) | 6 (6) | 1 (1)
DRY EYES (Eye disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
KERATITIS (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MELANOSIS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER SURGERY/PROCEDURE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARACENTRAL DEPRESSIONS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SJORGRENS SYNDROME (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SUBCONJUNCTIVAL HEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
XANTHELASMA (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL CRAMPS/PAIN (Gastrointestinal disorders) | 8 (8) | 1 (1) | 11 (11) | 5 (5)
ALTERED TASTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLACK STOOLS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 3 (3) | 5 (5) | 3 (3)
DIARRHEA/LOOSE STOOLS (Gastrointestinal disorders) | 8 (8) | 6 (6) | 5 (5) | 8 (8)
DIVERTICULITIS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
GERD (Gastrointestinal disorders) | 17 (17) | 2 (2) | 11 (11) | 5 (5)
GI FLU (Gastrointestinal disorders) | 13 (13) | 9 (9) | 12 (12) | 4 (4)
GI ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NAUSEA/VOMITING (Gastrointestinal disorders) | 11 (11) | 12 (12) | 11 (11) | 6 (6)
OCCLUDED/SWOLLEN SALIVARY GLAND (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL ULCERS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
OTHER INFECTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RECTAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ALOPECIA (General disorders) | 0 (0) | 1 (1) | 6 (6) | 0 (0)
ALTERED TASTE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
BURNING SENSATION (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CHILLS/SWEATS (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
DENTAL PAIN/INFECTION/ABSCESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 5 (5) | 8 (8) | 7 (7) | 3 (3)
HOARSENESS OF VOICE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLASHES (General disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
INJECTION SITE REACTION (General disorders) | 2 (2) | 3 (3) | 9 (9) | 0 (0)
INJURY (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
INSOMINA (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
INSOMNIA (General disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Other (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
SLEEP APNEA (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SORE TONGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNCOPY (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
TONGUE FISSURES (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VOICE HOARSENESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS/CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FATTY LIVER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 10 (10) | 2 (2) | 6 (6) | 2 (2)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
CANDIDIASIS (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
COMMON COLD (Infections and infestations) | 7 (7) | 2 (2) | 1 (1) | 1 (1)
COUGH (Infections and infestations) | 7 (7) | 0 (0) | 5 (5) | 4 (4)
DENTAL PAIN/INFECTION/ABSCESS (Infections and infestations) | 6 (6) | 2 (2) | 14 (14) | 9 (9)
DERMATALOGIC ERUPTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EARACHE/ INFECTION (Infections and infestations) | 12 (12) | 7 (7) | 5 (5) | 1 (1)
EYE INFECTION (Infections and infestations) | 5 (5) | 0 (0) | 5 (5) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
FLU /FLU LIKE SYMPTOMS (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
HERPES (Infections and infestations) | 5 (5) | 5 (5) | 7 (7) | 1 (1)
INFECTED FINGER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFECTED TOENAIL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHADENOPATHY/LYMPHADENITIS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
OTHER INFECTION (Infections and infestations) | 15 (15) | 7 (7) | 12 (12) | 9 (9)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
PROSTATE INFECTION/ENLARGEMENT (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
SINUS INFECTION (Infections and infestations) | 21 (21) | 13 (13) | 19 (19) | 11 (11)
SORE THROAT (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
STREP THROAT (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 131 (131) | 67 (67) | 146 (146) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 19 (19) | 6 (6) | 29 (29) | 8 (8)
Vaginal/Pelvic Infection (Infections and infestations) | 6 (6) | 5 (5) | 3 (3) | 2 (2)
Weight gain (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATALOGIC ERUPTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EXTREMITY SPRAIN/CRAMPS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 1 (1) | 2 (2)
INJURY (Injury, poisoning and procedural complications) | 9 (9) | 4 (4) | 12 (12) | 11 (11)
Joint Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anemia (Investigations) | 3 (3) | 4 (4) | 4 (4) | 2 (2)
ELEVATED CK AND ALDOLASE (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELEVATED CREATININE (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ELEVATED LIVER ENZYMES (Investigations) | 14 (14) | 1 (1) | 17 (17) | 5 (5)
HYPERCHOLESTEROLEMIA (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
HYPERGLYCEMIA (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
HYPERKALEMIA (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INCREASED ESR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LABORATORY ERROR (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOSIS/LEUKOPENIA (Investigations) | 5 (5) | 4 (4) | 2 (2) | 2 (2)
OTHER SURGERY/PROCEDURE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOSIS/THROMBOCYTOPENIA (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
VITAMIN B-12 DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 5 (5) | 3 (3)
EXTREMITY SPRAIN/CRAMPS (Musculoskeletal and connective tissue disorders) | 13 (13) | 7 (7) | 17 (17) | 4 (4)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
GOUT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEALED FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERNIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 66 (66) | 23 (23) | 57 (57) | 22 (22)
Joint Surgery/Procedure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mixed Connective Tissue Disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DERMATALOGIC ERUPTION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMP/NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2) | 9 (9) | 1 (1)
LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
SUBUNGUAL NEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THYROID ENLARGEMENT/NODULES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CHARCOT MARIE SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 7 (7) | 3 (3) | 8 (8) | 2 (2)
FACIAL DROOP (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 14 (14) | 8 (8) | 25 (25) | 6 (6)
MEMORY LOSS/CONFUSION (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
NEUROMA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 6 (6) | 0 (0) | 1 (1) | 1 (1)
NUMBNESS, DROOPING (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TREMORS (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ANXIETY/NERVOUSNESS/IRRITABILITY (Psychiatric disorders) | 0 (0) | 4 (4) | 4 (4) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 3 (3) | 4 (4) | 6 (6) | 3 (3)
METHADONE WITHDRAWAL (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL CALCULI (Renal and urinary disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
URINARY INCONTINENCE/FREQUENCY/URGENCY (Renal and urinary disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
ABNORMAL MENSES (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ATYPICAL PAP TEST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PROLAPSED UTERUS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATE INFECTION/ENLARGEMENT (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VAGINAL DISCHARGE/BLEEDING (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASTHMA/COPD (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NOSE BLEED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0)
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
BRITTLE FINGERNAILS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHILLS/SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DELAYED WOUND HEALING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DERMATALOGIC ERUPTION (Skin and subcutaneous tissue disorders) | 36 (36) | 16 (16) | 37 (37) | 14 (14)
INJURY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MELASMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NASAL IRRITATION/EROSION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ORAL ULCERS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
OTHER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER INFECTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PEELING SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PETECHIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLANTAR FASCITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
POOR WOUND HEALING (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUPRACLAVICULAR FAT PADS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Surgical and medical procedures) | 9 (9) | 0 (0) | 0 (0) | 1 (1)
DENTAL PAIN/INFECTION/ABSCESS (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
DERMATALOGIC ERUPTION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FRACTURE (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJURY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JOINT SURGERY/PROCEDURE (Surgical and medical procedures) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
OTHER SURGERY/PROCEDURE (Surgical and medical procedures) | 1 (1) | 2 (2) | 9 (9) | 8 (8)
CLAUDICATION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NOSE BLEED (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL VASCULAR DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less